CLINICAL TRIAL: NCT06010394
Title: Comparison of the Effectiveness of Exercise and Classical Massage in the Control of Edema in the Knee in Patients With Knee Osteoarthritis.
Brief Title: Control of Edema in the Knee in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar50
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Knee Osteoarthritis; Edema; Edema Leg
Keywords: massage
MeSH Terms: conditions — Osteoarthritis, Knee; Edema | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: classical physical therapy, exercise therapy, classical massage
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Active Comparator): commensal physiotherapy will be applied
  Interventions: Other: conventional physiotherapy
- exercise group (Experimental): exercises will be given
  Interventions: Other: conventional physiotherapy; Other: exercises for the knee area
- massage group (Experimental): massage will be done
  Interventions: Other: conventional physiotherapy; Other: payment oriented massage

INTERVENTIONS:
Other: conventional physiotherapy — ultrasound electrotherapy cold applications
Other: exercises for the knee area — range of motion exercises strengthening exercises exercises to reduce edema
  Arms: exercise group
Other: payment oriented massage — 10 / 15-minute massage treatments to reduce payment
  Arms: massage group

SUMMARY:
The aim of this study was to compare the effectiveness of exercise and classical massage in the control of knee edema in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
This study will be a prospective randomized controlled study. It is planned to include 75 patients with knee osteoarthritis in this study. It was categorized as osteoarthritis(OA) stages according to Kellgren-Lawrence criteria. Patients were randomly divided into three groups. the investigators first group is the control group (KG) and this group will receive classical physical therapy with ultrasound and subcutaneous electrical nerve stimulation. Exercise therapy will be applied to the second group in addition to the classical physical therapy applied to the KG. The third group will be given classical massage in addition to the classical physical therapy applied to the KG. The treatments to be applied to the patients will be 3 sessions per week and it is planned to continue for 4 weeks. Knee edema, pain severity, functional status and daily life activities will be measured at the beginning and in the 4th week of the patients. The data obtained will be analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 30-65
* Patients with a diagnosis of osteoarthritis in stage 2 and stage 3 according to Kellgren-Lawrence criteria(1) and also with measurable edema

Exclusion Criteria:

* Inability to continue treatment regularly
* situations that prevent you from doing the exercise
* inflammation that interferes with massage.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score | 4 weeks
  It is used to detect symptoms and restrictions in current work that individuals do in daily life. The test is collected under 2 main headings, consisting of 6 questions about the effect of symptoms and 8 sub-activities that question the status of the activity. The answer to each question in the test is scored between 0-5. The scores that the person gets from each question are added together and these scores are divided by 70 and multiplied by 100. High score means low quality of life.
Western Ontario and McMaster Universities Osteoarthritis Index | 4 weeks
  Pain, joint stiffness and functional status; Evaluated with the Arthritis Index of Western Ontario and McMaster Universities. The scale is a disease-specific, multidimensional, self-administered health status tool used in hip or knee osteoarthritis27. It consists of 24 questions on pain, stiffness and physical disability and is approximately 10 min. can be completed in Western Ontario and McMaster Universities Osteoarthritis Index consists of 24 questions under three sub-headings. Pain consists of 5 questions, stiffness 2 questions and function 17 questions. Each sub-parameter is scored between 0-4 points. Accordingly, it is classified as pain (0-20), stiffness (0-8) and function (0-68). A high score indicates poor health, a low score indicates good health.

CONTACTS AND LOCATIONS:
Overall Officials: Enver Deniz YILDIRIM, Study Chair — Uskudar University
Locations (1):
- Uskudar university, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maricar N, Callaghan MJ, Parkes MJ, Felson DT, O'Neill TW. Clinical assessment of effusion in knee osteoarthritis-A systematic review. Semin Arthritis Rheum. 2016 Apr;45(5):556-63. doi: 10.1016/j.semarthrit.2015.10.004. Epub 2015 Oct 22. PMID 26581486
- [Background] Hofmann S, Kramer J, Vakil-Adli A, Aigner N, Breitenseher M. Painful bone marrow edema of the knee: differential diagnosis and therapeutic concepts. Orthop Clin North Am. 2004 Jul;35(3):321-33, ix. doi: 10.1016/j.ocl.2004.04.005. PMID 15271540
- [Background] Molfetta L, Florian A, Saviola G, Frediani B. Bone Marrow Edema: pathogenetic features. Clin Ter. 2022 Sep-Oct;173(5):434-439. doi: 10.7417/CT.2022.2459. PMID 36155729
- [Background] Kan HS, Chan PK, Chiu KY, Yan CH, Yeung SS, Ng YL, Shiu KW, Ho T. Non-surgical treatment of knee osteoarthritis. Hong Kong Med J. 2019 Apr;25(2):127-133. doi: 10.12809/hkmj187600. Epub 2019 Mar 28. PMID 30919810